CLINICAL TRIAL: NCT00080067
Title: fMRI Study on Mechanism of Rhythm Perception and Generation
Brief Title: Rhythm Perception and Generation
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 040146; 04-N-0146
Record Dates: First submitted 2004-03-23; First posted 2004-03-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-23

CONDITIONS: Healthy
Keywords: Movement; Anticipation; Stimulation; Timing; Execution; Perception; Rhythm; Healthy Volunteer; HV

SUMMARY:
This study will examine how different brain areas are involved in the perception of rhythmic patterns and the performance of rhythmic movements. Patients with certain types of brain diseases, such as Parkinson's disease and some types of stroke, may have difficulty performing rhythmic movements, such as finger tapping.

Healthy, right-handed volunteers between 21 and 65 years of age may be eligible for this study. Candidates with visual, motor or hearing problems are excluded, as are musicians and pregnant women.

Participants will come to the National Institutes of Health (NIH) Clinical Center for up to six sessions of functional magnetic resonance imaging (fMRI) scanning. MRI uses a strong magnetic field and radio waves to obtain images of body organs and tissues. The scanner is a metal cylinder surrounded by a magnetic field. During the MRI, the subject lies still for up to 20 minutes at a time on a table in the cylinder and wears earplugs to muffle loud knocking noises that occur with the electrical switching of the magnetic fields. He or she can communicate with the MRI staff through a microphone at all times during the procedure.

For fMRI, images are obtained while the subject performs a task, such as hearing sounds or moving a finger. The machine detects changes in brain movement that are involved in performing the task. The tasks are explained, and subjects can practice them before entering the scanner.

DETAILED DESCRIPTION:
Objective

Rhythmic movements, such as finger tapping, are relatively simple. However, many brain areas including motor, somatosensory, premotor and prefrontal cortex, supplementary motor area, basal ganglia, cerebellum, etc. have been reported to be activated during rhythmic movements. Patients with lesions located in the extrapyramidal or cerebellar system, such as patients with Parkinson's disease, cerebellar ataxia or stroke with a lesion in these systems, have difficulties in performing rhythmic movements. Timing deficits after basal ganglia or cerebellar damage could also be due to abnormalities in interconnecting cortical systems commonly associated with these processes. Few studies have examined involvement of cerebral cortex in time perception.

The purpose of this study is to detect the brain areas associated with three hypothesized processes associated with rhythm perception and generation: (1) perception of external rhythmic stimulation, (2) internal rhythm generation and (3) execution of rhythmic movement. To investigate whether the process of rhythm perception is common across sensory modalities, we will use auditory and visual stimulation.

Study population

This research will be conducted using normal adult volunteers.

Design

Using functional magnetic resonance imaging, we will examine the brain activity of subjects while they will hear or watch rhythmic stimulation and press buttons rhythmically with their fingers. A series of experiments will be designed to demonstrate the hypothesized three processes separately.

Outcome measures

The brain activity correlated with experimental conditions and behavioral data (the timing error of button press to the corresponding rhythmic stimulation) will be collected and analyzed by using statistical parametric mapping (SPM).

The findings we expect to obtain with this experiment will contribute to basic knowledge for better understanding of the pathophysiology of the disturbance of perception and generation of rhythm in patients with neurological disorders, and give theoretical background for repetitive, rhythmically patterned movement training in neurorehabilitation.

ELIGIBILITY:
* INCLUSION CRITERIA:

Fifty healthy, right-handed adult (aged between 21 to 65 years old) volunteers will be recruited from people who are registered as HMCS normal volunteers. All subjects participating in MR studies should have a valid Clinical Center Medical Record Number.

Female subjects of childbearing potential will have a pregnancy test and a specific interview prior to the study to ensure that pregnant subjects will not participate in the study.

EXCLUSION CRITERIA:

Subjects with implanted devices such as pacemakers, medication pumps or defibrillators, metal in the cranium except mouth, intracardiac lines, history of shrapnel injury or any other condition/device that may be contraindicated or prevent the acquisition of MRI.

Pregnant female. A pregnancy test will be performed within 24 hours preceding each MRI and if the result is positive, that subject will not be studied.

Subjects with claustrophobia

Subjects with any visual, motor or hearing difficulties

Musicians

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2004-03-22; Study Completion 2009-02-23

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Artieda J, Pastor MA, Lacruz F, Obeso JA. Temporal discrimination is abnormal in Parkinson's disease. Brain. 1992 Feb;115 Pt 1:199-210. doi: 10.1093/brain/115.1.199. PMID 1559154
- [Background] Aschersleben G. Temporal control of movements in sensorimotor synchronization. Brain Cogn. 2002 Feb;48(1):66-79. doi: 10.1006/brcg.2001.1304. PMID 11812033
- [Background] Asanuma H, Keller A. Neuronal mechanisms of motor learning in mammals. Neuroreport. 1991 May;2(5):217-24. doi: 10.1097/00001756-199105000-00001. PMID 1912451